CLINICAL TRIAL: NCT02478216
Title: The Effect of Remote Ischemic Preconditioning on Postoperative Cognitive Dysfunction in Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Seong-Hyop Kim, Professor, Konkuk University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KUH1160078
Record Dates: First submitted 2015-04-20; First posted 2015-06-23 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- C group (No Intervention): Remote ischemic preconditioning will not be applied
- R group (Experimental): Remote ischemic preconditioning will be applied.
  Interventions: Procedure: Remote ischemic preconditioning

INTERVENTIONS:
Procedure: Remote ischemic preconditioning — The tourniquet was applied at the opposite site from operation thigh in the both groups. The thigh was covered with blanket to conceal the tourniquet inflation and deflation. A total of 3 cycles of tourniquet inflation for 5 minutes with 2 × systemic systolic arterial blood pressure of arrival at operation room and deflation were performed.
  Arms: R group

SUMMARY:
The patients were allocated randomly to receive remote preconditioning group (RIPC group, R) or not (Control group, C) using sealed envelopes with the options inside the sealed envelope of R and C before anaesthesia induction. The registered nurse who did not participate in patient care and was blind to the study performed the all randomization process. All medical staffs who involved the patient care were blind to the study. All data were collected by trained observers who were blind to the study and did not participate in patient care

DETAILED DESCRIPTION:
RIPC was performed just after anesthesia induction and before the tourniquet application for the operation site. The tourniquet was applied at the opposite site of thigh in the both groups. The thigh was covered with blanket to conceal the tourniquet inflation and deflation. For R group, 3 cycles of tourniquet inflation for 5 minutes with 2 × systemic systolic arterial blood pressure of arrival at operation room and deflation were performed. For C group, the tourniquet was applied with same manner for R group except inflation pressure of 0 mmHg. The tourniquet pressure according to the randomization was set by the registered nurse who participated in the patients' allocation. The monitor of tourniquet pressure was sealed for blindness.

ELIGIBILITY:
Inclusion Criteria:

* patient who was planned to undergo total knee replacement surgery

Exclusion Criteria:

* emergency operation
* underlying cerebrovascular disease
* underlying peripheral vascular disease

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Incidence of cerebral desaturation | during operation time (an expected average of 2 hours)
  cerebral saturation will be assessed by using near infrared spectroscopy

SECONDARY OUTCOMES:
Incidence of postoperative delirium | up to postoperative 7 days
  postoperative delirium will be assessed by using CAM method.

CONTACTS AND LOCATIONS:
Overall Officials: Seong-Hyop Kim, M.D,Ph.D, Principal Investigator — Konkuk University Medical Center
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea